CLINICAL TRIAL: NCT02534129
Title: Topical Use of a Silibin-based Cream, Difinsa53™, to Prevent Radiation Dermatitis in Patients With Breast Cancer: A Prospective Study
Brief Title: Topical Use of Difinsa53™ to Prevent Radiation Dermatitis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient dermatitis was seen in the controls to allow any determination of protection by Difinsa53
Sponsor: ProTechSure Scientific, Inc. (Industry)
Collaborators: Poudre Valley Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ProTechSure 001
Record Dates: First submitted 2015-08-19; First posted 2015-08-27 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Radiodermatitis
Keywords: breast cancer; radiation; dermatitis
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms; Dermatitis | interventions — dimethicone; Petrolatum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Radiation field is divided into two sections, one treated with Difinsa53 and the other with Aquaphor
  Interventions: Drug: Difinsa53; Drug: Aquaphor

INTERVENTIONS:
Drug: Difinsa53 — Difinsa53 cream is applied to one half of radiation field
  Other Names: Dimethicone
Drug: Aquaphor — Aquaphor is applied to one half of radiation field
  Other Names: petrolatum

SUMMARY:
Phase II trial of the silibin containing cream, Difinsa53 to determine efficacy in delaying, ameliorating, or preventing radiation dermatitis in patients with breast cancer undergoing whole breast radiation.

DETAILED DESCRIPTION:
The proposed study seeks to evaluate the efficacy of DIFINISA53™, a safe silibin-based skin cream, on preventing radiation dermatitis (RD) when compared to an over the counter ointment, Aquaphor, in women undergoing radiation therapy for breast cancer following lumpectomy or mastectomy surgery. Presently there is no known fully effective topical protectant from RD and there is no consensus among radiation oncologists on how best to treat RD. This study seeks to identify a more effective option for patients receiving radiation therapy. Each participant will apply the DIFINISA53™ cream to one area of the treated skin and Aquaphor to another area of treated skin. Skin reactions will be evaluated using medical professional assessment, participant assessment, and photographic assessment by a third party.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years and older
* Pathologic diagnosis of breast cancer requiring radiation therapy to whole breast
* Able to apply lotion to treatment area at least twice daily during radiation course
* All surgical sites healed
* No evidence of infection
* No history of sensitivity to any component in Aquaphor or Difensa53

Exclusion Criteria:

* Prior history of radiation therapy (RT) to that site
* Known dermatologic conditions affecting skin in radiation port
* Concurrent chemotherapy
* Skin infection in radiation port
* History of sensitivity to Aquaphor or Difensa53 component

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Petit, MD, Principal Investigator — UC Health, Poudre Valley Hospital
Locations (1):
- Poudre Valley Health System, Fort Collins, Colorado, United States

REFERENCES:
- [Background] McQuestion M. Evidence-based skin care management in radiation therapy: clinical update. Semin Oncol Nurs. 2011 May;27(2):e1-17. doi: 10.1016/j.soncn.2011.02.009. PMID 21514477
- [Background] Becker-Schiebe M, Mengs U, Schaefer M, Bulitta M, Hoffmann W. Topical use of a silymarin-based preparation to prevent radiodermatitis : results of a prospective study in breast cancer patients. Strahlenther Onkol. 2011 Aug;187(8):485-91. doi: 10.1007/s00066-011-2204-z. Epub 2011 Jul 22. PMID 21786113

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 patients were entered, each of whom had a single radiation port divided into two fields. One received aquaphor protection and the other received Difinsa53 protection.
Units Other Than Participants: Radiation fields
Groups:
- Aquaphor: This radiation field treated with aquaphor
- Difinsa53: This radiation field treated with Difinsa53
Period: Overall Study
Arm/Group | Aquaphor | Difinsa53
Started | 13; 13 Radiation fields | 13; 13 Radiation fields
Completed | 13; 13 Radiation fields | 13; 13 Radiation fields
Not Completed | 0; 0 Radiation fields | 0; 0 Radiation fields

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of 13 breast cancer patients receiving radiation to a breast. Each breast was divided into two radiation fields, one defined as the Difinsa53 arm and the other as the Aquaphor Arm. Thus each participant contributed data from two fields.
Groups:
- Difinsa53 and Aquaphor Arms: Radiation field is divided into two sections, one treated with Difinsa53 and the other with Aquaphor
  Difinsa53: Difinsa53 cream is applied to one half of radiation field
  Aquaphor: Aquaphor is applied to one half of radiation field
Arm/Group | Difinsa53 and Aquaphor Arms
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Participants: Female | 13
  Participants: Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Radiation Dermatitis as Determined by Radiation Therapy Oncology Group (RTOG) Acute Radiation Morbidity Scoring Criteria
Description: A blinded observer will quantify degree of dermatitis assigning each half of the radiation field a score from 0 to 4. 0 represents no dermatitis and 4 is severe dermatitis using the RTOG scoring criteria.
Time Frame: 8 weeks
Population: All patients were analyzed by blinded observor
Measure: Median (Full Range); unit: units on a scale
Groups:
- Difinsa 53 Arm: Radiation field is divided into two sections, one treated with Difinsa53 and the other with Aquaphor
  Difinsa53: Difinsa53 cream is applied to one half of radiation field
- Aquaphor Arm: Radiation field is divided into two sections, one treated with Difinsa53 and the other with Aquaphor
  Aquaphor: Aquaphor is applied to one half of radiation field
Arm/Group | Difinsa 53 Arm | Aquaphor Arm
Number analyzed (Participants) | 13 | 13
units on a scale | 0 [0 to 1] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: Data were collected over 12 weeks for each arm.
Groups:
- Difinsa53 Arm: Radiation field is divided into two sections, one treated with Difinsa53 and the other with Aquaphor
  Difinsa53: Difinsa53 cream is applied to one half of radiation field
Arm/Group | Difinsa53 Arm | Aquaphor Arm
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
This trial was terminated early, based on minimal radiation dermatitis (scores of 0-1 only in most fields evaluated) that precluded any meaningful analysis of any differing effect in the two treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No